CLINICAL TRIAL: NCT04228484
Title: Beta Cell Responsiveness to Glucose-dependent Insulinotropic Polypeptide Following Near-normalisation of Plasma Glucose in Overweight Patients With Type 2 Diabetes
Brief Title: The Insulin Response to the Gut Hormone GIP After Near-normalisation of Plasma Glucose in Patients With Type 2 Diabetes
Acronym: GA-16
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, MD, PhD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-19069850
Record Dates: First submitted 2020-01-07; First posted 2020-01-14 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Type2 Diabetes
Keywords: Type 2 Diabetes,; Incretin Effect; GIP; Glucose-dependent Insulinotropic Polypeptide
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo infusion
  Interventions: Other: Placebo
- GIP receptor antagonization (Active Comparator): GIP(3-30)NH2 infusion
  Interventions: Other: GIP receptor antagonization

INTERVENTIONS:
Other: Placebo — Placebo infusion
  Arms: Placebo
Other: GIP receptor antagonization — GIP(3-30)NH2 infusion
  Arms: GIP receptor antagonization

SUMMARY:
The investigators hypothesise that the insulinotropic effect of endogenous GIP is improvable in patients with type 2 diabetes after three weeks of near-normalisation of plasma glucose. To test this hypothesis, a randomised, placebo-controlled, double-blinded, crossover study employing a GIP receptor antagonist, will be carried out.

Fifteen overweight (body mass index (BMI) > 25 kg/m2) dysregulated (HbA1c >/= 59 mmol/mol and treatment with metformin or >53 mmol/mol and treatment with metformin + add/on) patients with type 2 diabetes will attend two experimental days followed by a three-week-four-week period of plasma glucose near-normalisation (achieved by standard treatment of type 2-diabetes), followed by another two experimental days. On experimental days, patients will receive an infusion of GIP receptor antagonist or placebo during a 75 g oral glucose tolerance test. The primary endpoint is changes in levels of C-peptide divided by changes in levels of plasma glucose and secondary endpoints include changes in circulating levels of C-peptide, insulin, glucose, GIP, glucagon-like peptide 1 (GLP-1), glucagon and markers of bone turnover as well as indices of beta cell function. Furthermore, gastric emptying rate will be assessed.

DETAILED DESCRIPTION:
Glucose-dependent insulinotropic polypeptide (GIP) exerts a strong insulinotropic effect in healthy individuals following meal ingestion. Studies in patients with type 2 diabetes have shown that the insulinotropic effect of exogenous GIP is severely reduced and recent data from the investigators' group suggest that the insulinotropic effect of endogenous GIP is compromised too. Interestingly, after near-normalisation of plasma glucose in patients with type 2 diabetes (continuing metformin and by using empagliflozin + intensive insulin treatment), the insulinotropic effect of exogenous GIP can be restored. The investigators have previously observed a similar restoration of the beta cell secretory response to exogenous GIP after therapy with DPP-4 inhibitors, the effects of which rely on preservation of incretins.

The investigators hypothesise that the insulinotropic effect of endogenous GIP is improvable in patients with type 2 diabetes after three weeks-four weeks of near-normalisation of plasma glucose. To test this hypothesis, a randomised, placebo-controlled, double-blinded, crossover study employing a GIP receptor antagonist, will be carried out.

Fifteen overweight (body mass index (BMI) > 25 kg/m2) dysregulated (HbA1c >/= 59 mmol/mol and treatment with metformin or >53 mmol/mol and treatment with metformin + add/on) patients with type 2 diabetes will attend two experimental days followed by a three-week/four-week period of plasma glucose near-normalisation (achieved by standard treatment of type 2-diabetes), followed by another two experimental days. On experimental days, patients will receive an infusion of GIP receptor antagonist or placebo during a 75 g oral glucose tolerance test. The primary endpoint is changes in levels of C-peptide divided by changes in levels of plasma glucose and secondary endpoints include changes in circulating levels of C-peptide, insulin, glucose, GIP, glucagon-like peptide 1 (GLP-1), glucagon and markers of bone turnover as well as indices of beta cell function. Furthermore, gastric emptying rate will be assessed.

Glucose-lowering drugs based on the effects of another incretin hormone, GLP-1, are successfully being used in the treatment of type 2 diabetes. However, due to the reduced insulinotropic effect of GIP in patients with inadequately controlled type 2 diabetes, treatments based on GIP receptor activation are not on the market. Recently however, a dual GLP-1/GIP receptor agonist has shown promising phase II results. The importance of GIP receptor engagement for the efficacy of these compounds remains to be shown. The present project will answer to what extent the insulinotropic effect of endogenous GIP in patients with type 2 diabetes can be restored following near-normalisation of plasma glucose and thus, provide important perspectives on how to further advance the development of GIP-based therapeutics.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. Metformin treatment
3. Haemoglobin A1c (HbA1c) I. >/= 59 mmol/mol in case the diabetes treatment is only metformin II. 53-75 mmol/mol in case the diabetes treatment is metformin and add-on therapy
4. Body Mass Index (BMI) > 25 kg/m2
5. Age > 18 years
6. Caucasian
7. Normal haemoglobin levels

Exclusion Criteria:

1. Treatment with GLP-1-receptor agonist
2. Any treatment that cannot be paused for 12 hours
3. Diabetes duration more than 20 years
4. Weekly alcohol intake of more than 14 units for men or 7 units for women of alcohol (of 12 g) or narcotics abuse
5. Liver disease
6. Kidney disease (estimated glomerular filtration rate, eGFR < 60 ml/min/1,73 m2)
7. Unusual dietary preferences or planned weight loss within the duration of the study
8. Any other condition that in the opinion of the responsible investigators is disqualifying.
9. For women I. Current or planned pregnancy for the duration of the study II. Positive pregnancy test at the screening or any of the experimental days III. Women who are currently breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change in [plasma C-peptide] / [plasma glucose] after near-normalisation of plasma glucose | Assessed multiple times on each of the four study days
  The primary endpoint is beta cell sensitivity to glucose as assessed by the C-peptide response to a 75 g-oral glucose tolerance test (OGTT) (as assessed by baseline-subtracted area under the curve (bsAUC)) divided by levels of plasma glucose (as assessed by bsAUC) during GIP(3-30)NH2 infusion compared to placebo before and after near-normalisation of plasma glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, Professor, MD, Principal Investigator — Director of Center for Clinical Metabolic Research, Gentofte Hospital
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gasbjerg LS, Helsted MM, Hartmann B, Jensen MH, Gabe MBN, Sparre-Ulrich AH, Veedfald S, Stensen S, Lanng AR, Bergmann NC, Christensen MB, Vilsboll T, Holst JJ, Rosenkilde MM, Knop FK. Separate and Combined Glucometabolic Effects of Endogenous Glucose-Dependent Insulinotropic Polypeptide and Glucagon-like Peptide 1 in Healthy Individuals. Diabetes. 2019 May;68(5):906-917. doi: 10.2337/db18-1123. Epub 2019 Jan 9. PMID 30626611